CLINICAL TRIAL: NCT03140904
Title: Reducing the Frequency of Follow up and Task Sharing in the Treatment of Uncomplicated Severe Acute Malnutrition: an Evaluation of Monthly Visits and Home-based Surveillance for Access-limited and High-burden Settings
Brief Title: Reducing the Frequency of Follow up and Task Sharing in the Treatment of Uncomplicated Severe Acute Malnutrition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Epicentre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Reduced follow-up
Record Dates: First submitted 2017-04-28; First posted 2017-05-04 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Severe Acute Malnutrition
MeSH Terms: conditions — Severe Acute Malnutrition

STUDY DESIGN:
Intervention Model Description: 1. Standard weekly visits at the outpatient therapeutic feeding center until discharge
  2. Monthly visits at the outpatient therapeutic feeding center with caregiver support for home-based surveillance, with visits scheduled at weeks 4, 8, 10 and 12 until discharge.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard weekly visits (Other): Standard weekly visits at the outpatient therapeutic feeding center until discharge
  Interventions: Other: Standard weekly visits
- Monthly visits (Other): Monthly visits at the outpatient therapeutic feeding center with caregiver support for home-based surveillance, with visits scheduled at weeks 4, 8, 10 and 12 until discharge
  Interventions: Other: Monthly visits

INTERVENTIONS:
Other: Standard weekly visits — Distribution of the therapeutic feeding rations, as well as medical and anthropometric surveillance, will take place on a weekly basis at the outpatient therapeutic feeding center according to the random assignment of the site, until discharge
  Arms: Standard weekly visits
Other: Monthly visits — Distribution of the therapeutic feeding rations, as well as medical and anthropometric surveillance, will take place on a monthly basis at the outpatient therapeutic feeding center according to the random assignment of the site, until discharge
  Arms: Monthly visits

SUMMARY:
This study will be conducted as a stratified cluster randomized trial. The unit of randomization will be the outpatient therapeutic feeding center. The 10 health centers will be stratified by size, and centers within a stratum will be randomized in a 1:1 ratio to one of two schedules of treatment: (1) standard weekly visits or (2) monthly visits with support for home-based surveillance.

DETAILED DESCRIPTION:
This study will be conducted as a stratified cluster randomized trial of a monthly schedule of follow up in the treatment of uncomplicated SAM among children aged 6 to 59 months. The unit of randomization will be the outpatient therapeutic feeding center. The 10 health centers supported by International Medical Corps UK (IMC-UK) will be stratified by size (± 1000 admissions per site per year), and centers within a stratum will be randomized in a 1:1 ratio to one of two schedules of treatment: (1) standard weekly visits or (2) monthly visits with support for home-based surveillance.

Distribution of the therapeutic feeding rations, as well as medical and anthropometric surveillance, will take place on a weekly or monthly basis until discharge according to the random assignment of the site. Caregivers in the monthly visit group will receive additional instruction at admission regarding home-based MUAC measurement and clinical surveillance.

Regardless of intervention assignment, all children with uncomplicated SAM will receive standard medical care on admission as per national guidelines, and a home visit 2 months following discharge from the nutritional program. Additional data collection, including coverage assessment and economic costing analysis will be used to address the secondary objectives related to the evaluation of coverage and cost-effectiveness, respectively.

ELIGIBILITY:
Inclusion Criteria:

* age from 6 to 59 months
* MUAC < 115 mm and/or grade 1-2 edema
* Absence of current illness requiring inpatient care

Exclusion Criteria:

* History of allergy to peanuts
* Any other condition in which, in the judgment of the Field Investigator, would interfere with or serves as a contraindication to protocol adherence or the ability to give informed consent

Ages: 6 Weeks to 59 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3945 (Actual)
Dates: Start 2018-01-23 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-04-27 (Actual)

PRIMARY OUTCOMES:
Nutritional recovery | Minimum length of stay is 8 weeks
  Defined by being free from medical complications, MUAC > 125 mm, and no edema for 2 weeks if admitted with edema

SECONDARY OUTCOMES:
Hospitalization | within 2 months
  Hospitalization, defined as referral to inpatient care for weight/edema change, or failed appetite test, clinical complication necessitating inpatient care
Daily weight gain (g / kg / day) among recovered children | within 2 months
  difference in weight (g)
Defaulting | within 2 months
  3 missed scheduled facility visits in the weekly follow-up group and 1 missed scheduled facility visit in the monthly follow-up group
Relapse | Within 2 months
  Maternal report of admission to any therapeutic feeding program

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca GRAIS, Study Director — Epicentre
Locations (1):
- Sokoto State Nutrition Centre, Sokoto, Nigeria

IPD SHARING:
Plan to Share IPD: Undecided
Subject to individual data sharing agreements

REFERENCES:
- [Derived] Ali NB, Hitchings MD, Berthe F, Aruna P, Shehu I, Nanama S, Steve-Edemba C, Grais RF, Isanaka S. Effect of caregiver training on knowledge and confidence of at-home clinical and anthropometric surveillance of children with uncomplicated severe acute malnutrition: analysis of a cross-over cluster randomised trial in Sokoto, Nigeria. BMJ Glob Health. 2025 Oct 6;10(10):e018559. doi: 10.1136/bmjgh-2024-018559. PMID 41057203
- [Derived] Menzies NA, Berthe F, Hitchings M, Aruna P, Hamza MA, Nanama S, Steve-Edemba C, Shehu I, Grais RF, Isanaka S. Cost-effectiveness of monthly follow-up for the treatment of uncomplicated severe acute malnutrition: An economic evaluation of a randomized controlled trial. PLOS Glob Public Health. 2022 Dec 9;2(12):e0001189. doi: 10.1371/journal.pgph.0001189. eCollection 2022. PMID 36962786
- [Derived] Hitchings MDT, Berthe F, Aruna P, Shehu I, Hamza MA, Nanama S, Steve-Edemba C, Grais RF, Isanaka S. Effectiveness of a monthly schedule of follow-up for the treatment of uncomplicated severe acute malnutrition in Sokoto, Nigeria: A cluster randomized crossover trial. PLoS Med. 2022 Mar 1;19(3):e1003923. doi: 10.1371/journal.pmed.1003923. eCollection 2022 Mar. PMID 35231024
- [Derived] Isanaka S, Hedt-Gauthier BL, Salou H, Berthe F, Grais RF, Allen BGS. Active and adaptive case finding to estimate therapeutic program coverage for severe acute malnutrition: a capture-recapture study. BMC Health Serv Res. 2019 Dec 16;19(1):967. doi: 10.1186/s12913-019-4791-9. PMID 31842870